CLINICAL TRIAL: NCT04849104
Title: Cohort Study of Airway Microecology and the Pathogenesis and Evolution of Chronic Obstructive Pulmonary Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Other Study IDs: COPD-BALF2021
Record Dates: First submitted 2021-04-08; First posted 2021-04-19 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 60ml bronchoalveolar lavage fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- COPD high-risk patients: age <70 years old, long-term smoker (≥10 pack years), CT without macroscopic airway abnormalities and/or mild or moderate emphysema, air retention or bronchial thickening, normal lung function
- Early-stage COPD patients: those who are younger than 70 years old, long-term smokers (≥10 pack years) and have any of the following abnormalities:
  1. Forced expiratory volume in the first second/forced vital capacity (FEV1/FVC) <lower limit of normal value (LLN, 80%);
  2. CT abnormalities: abnormal airway and/or emphysema, air retention or bronchial wall thickening;
  3. FEV1 drops rapidly (≥60 mL/year);
- patients with mild to moderate COPD: Patients with mild to moderate COPD: age <75 years, FEV1/FVC<70%, FEV1 predicted value ≥50%

SUMMARY:
This study will last for 5 years (2021.2.25-2025.12.31). 210 patients (70 cases in each group) will be enrolled in this study. Eight centers in China will participate in the study. The patients will be treated with bronchoscopy alveolar lavage, and 60 ml of bronchoalveolar lavage fluid will be collected for the next-generation sequencing of airway microorganisms. The patients will be followed up for 4 years to observe the changes of lung function, Fractional exhaled nitric oxide (FENO) and clinical symptoms.

DETAILED DESCRIPTION:
1. Research purposes:

   The main purpose: to detect the relationship between the changes in the airway microecology and the activation of macrophages, as well as the progression and heterogeneity of the early disease of COPD in patients with early COPD.

   The basis of the question:

   The current study found that the number of patients with COPD in my country is close to 100 million, and the number of deaths due to COPD every year ranks third among the deaths of each single disease in my country. However, the research on the pathogenesis of COPD has been slow and there is still no breakthrough. The results of research have brought innovations to the treatment of chronic obstructive pulmonary disease. The study found that the airway microecology has undergone significant changes in patients with moderate to severe COPD, but whether the airway microecology changes in the early COPD? If it changes, the airway microecology changes slowly in the early stage. What is the role in the evolution of obstructive lung disease? There is no relevant research report. This study intends to collect bronchoalveolar lavage fluid to detect the airway microecology and the activation of macrophages, and observe the changes in the airway microecology and the activation of macrophages in early COPD patients, as well as the early COPD Correlation between disease progression and heterogeneity.
2. Research design:

   Planned number of cases: 70 cases of COPD high-risk patients/early COPD/mild-moderate COPD patients, a total of 210 cases. The main center plans to enroll 28 cases, each sub-center plans to enroll 26 cases, and each center enters the group competitively.
3. Clinical trial process:

   3.1 Sign informed consent and collect relevant clinical data; for patients who are clearly diagnosed as COPD, the treatment plan formulated in the "Global Initiative for the Diagnosis, Treatment and Prevention of COPD" (the 2021 version of the GOLD Guidelines) Carry out standardized treatment.

   3.2 Under local anesthesia, perform bronchoalveolar lavage and recover bronchoalveolar lavage fluid;

   3.3 The recovered bronchoalveolar lavage fluid is divided into two parts. One part uses 16SrRNA high-throughput sequencing to detect the characteristics of the airway microecological composition of early COPD patients, and analyze the heterogeneity of the microecological composition of individual samples of early COPD patients. The other part of the specimen was centrifuged to separate the bronchoalveolar lavage fluid supernatant and cells.

   3.4 The cells in the bronchoalveolar lavage fluid were separated from macrophages by differential adhesion method, and M1 (CD68+CD80+CD86+CD163-CD206-) and M2 (CD68+CD80-CD86-) were detected by flow cytometry. CD163+CD206+) ratio; 3.5 The above-mentioned patients and healthy volunteers were followed up for 4 times in 4 years, and the changes in relevant clinical data were recorded. Primary endpoint: changes in lung function in high-risk patients with COPD/early COPD and mild-to-moderate COPD within 48 months; secondary endpoint: patients with high-risk COPD/early COPD patients and mild Changes in clinical symptoms in patients with moderate chronic obstructive pulmonary disease within 48 months. Analyze the correlation between airway microecological changes, the heterogeneity of microecological composition ratio, macrophage activation and the disease progression and heterogeneity of early COPD patients.

   (Remarks: If the subject has an acute exacerbation of chronic obstructive pulmonary disease at the time of follow-up, he will be treated according to the diagnosis and treatment standards, and the visit task at this node will be completed after the acute exacerbation is relieved for 1 month. )
4. quality assurance of clinical trial data

   The quality control of this clinical trial is under the control and control of the 9th People's Hospital Affiliated to the Medical College of Shanghai Jiaotong University. The research work is carried out in accordance with GCP, SOP and quality control requirements, the clinical research plan is formulated, and GCP training is conducted for the relevant researchers participating in the test.

   4.1 The plan before the trial is started shall be submitted to the ethics committee of the Ninth People's Hospital Affiliated to the Medical College of Shanghai Jiaotong University for approval;

   4.2 According to the GCP guidelines, necessary steps should be taken in the design and implementation stage of the study to ensure the accuracy, consistency, integrity and credibility of the collected data;

   4.3 The participants will conduct the test in strict accordance with the GCP standard in China, collect and record the contents in the case report form truthfully, carefully and in detail according to the SOP of clinical trial standard, and verify the contents to ensure the reliability of the data;

   4.4 The researchers fill in the information required by the program into the case report form (CRF), and the supervisor will verify that the information is complete and accurate, and guide the staff of the research center to make necessary corrections and supplements;

   4.5 All instruments, equipment, reagents, standard products, etc. used in various inspection items in clinical trials shall have strict quality standards and ensure that they work under normal conditions;

   4.6 The statistical problems in the test plan shall be submitted to the statistical experts for examination and verification;

   4.7 During the trial, researchers monitored the research process, informed consent, the correctness and completeness of data in case report form (CRF).
5. record, preservation, sharing agreement and declaration of conflict of interest of research materials

   According to GCP principle, the researcher shall keep all the detailed original documents of the subjects, and record the contents of the test process, drug use, laboratory examination data, safety data and efficacy evaluation in the case report form. The recorded data shall be complete, timely and clear. The case report form, original documents, medical records, etc. shall be clear, detailed and easily recognized by the personnel participating in this clinical trial.

   The key investigator must sign at least the selected confirmation page and completion page of the case report form to verify the accuracy and integrity of all data.

   The case report form and original documents can only be modified by the investigator. No modification to the case report form and original document shall be allowed to smear out the original data. The correct method of modification is to mark single line on the original data, then write the modified data next to the original data, and sign the date and the abbreviation of the modified personnel.

   The test data shall be kept for 10 years after the end of the test. However, if required by the current regulations or in agreements with the sponsor, the information should be kept for a longer period of time.

   The research results are shared by the contribution ranking of each center. There is no conflict of interest in each research center.
6. statistical treatment scheme

   6.1 filling in the case report form (CRF) The investigator should complete the filling of case report form in time, modify it according to the correct modification method, and the completed case report form shall be reviewed and signed by the main researchers.

   6.2 statistical analysis method and statistical description

   6.2.1 Treatment of missing value of main efficacy index data: when some subjects lack a major efficacy data, the method of filling deficiency is determined from the statistical and professional perspective. If the case is missing, the data of the previous measurement shall be transferred.

   6.2.2 Case analysis of incomplete test: the reasons for exfoliation should be analyzed one by one.

   6.2.3 Descriptive statistics: mean, standard deviation, maximum value, minimum value, median, confidence interval, frequency (composition ratio), etc.

   6.3 Statistical expression

   6.3.1 The report mainly uses tables to show that the tables are self-evident, that is, they have table questions, table notes and examples.

   6.3.2 The results of repeated measurement data are expressed in tables and statistical charts are attached to increase readability.

   6.4 statistical software

   SAS 9.1.3 and Das for clinical trial 3.0 software were used to analyze the software simultaneously, and the results were confirmed.
7. modification and interim analysis in the course of the test

Once the research plan has been discussed by the research group and reviewed by the ethics committee, it is not allowed to change at will; before the modification is implemented, the researcher must report the content and reason of the modification to the ethics committee of clinical trial for approval, and then carry out the research according to the modified scheme.

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to communicate orally or in writing and sign an informed consent form;
2. Age from 18 to 70 years (the age of patients with mild to moderate COPD <75 years), regardless of gender;
3. Meet the above-mentioned early diagnosis criteria for high-risk patients with COPD/early-stage COPD/mild to moderate COPD.

Exclusion Criteria:

1. Patients suffering from any of the following diseases: active tuberculosis, severe bronchiectasis, lung abscess, aspiration pneumonia, lung tumor, non-infectious interstitial lung disease, pulmonary edema, atelectasis, pneumothorax, pleural effusion , Pulmonary embolism, pulmonary eosinophilic infiltration, and pulmonary vasculitis;
2. Patients with a history of tumors or patients with current tumors;
3. The patient has severe renal impairment: creatinine clearance rate <30ml/min/1.73m2 or serum creatinine>265μmol/L (>3mg/dL);
4. Patients suffering from liver disease or severe liver damage: ALT, AST> 2 times the upper limit of normal;
5. pregnancy;
6. Severe COPD, FEV1 predicted value ≤50%;
7. Severe heart disease, such as coronary heart disease, heart failure, etc.;
8. Severe coagulopathy: INR>1.4, PTT>40s, PLT<150x103 cells
9. Bronchial Asthma;
10. Severe alcoholism;
11. diabetes;
12. Have used antibiotics within two months,
13. Used systemic and local hormones;
14. Cannot sign the informed consent form;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatient or hospitalized patient
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2021-02-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Forced vital capacity(FVC) | 0， 12，24，36，48months
  The change of FVC at each time node
Forced expiratory volume in the first second(FEV1) | 0， 12，24，36，48months
  The change of FEV1 at each time node
Forced expiratory rate in the first second (FEV1%=FEV1/FVC) | 0， 12，24，36，48months
  The change of FEV1% at each time node
Exhaled nitric oxide (FENO) | 0， 12，24，36，48months
  The change of FENO at each time node

SECONDARY OUTCOMES:
breathlessness measurement using the modified British Medical Research Council (mMRC) | 0， 12， 24， 36， 48months
  The change of mMRC at each time node
COPD assessment test (CAT) | 0， 12， 24， 36， 48months
  The change of CAT at each time node

CONTACTS AND LOCATIONS:
Overall Officials: Weining Xiong, doctor, Study Chair — Shanghai Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Ninth People's Hospital Affiliated to Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang C, Xu J, Yang L, Xu Y, Zhang X, Bai C, Kang J, Ran P, Shen H, Wen F, Huang K, Yao W, Sun T, Shan G, Yang T, Lin Y, Wu S, Zhu J, Wang R, Shi Z, Zhao J, Ye X, Song Y, Wang Q, Zhou Y, Ding L, Yang T, Chen Y, Guo Y, Xiao F, Lu Y, Peng X, Zhang B, Xiao D, Chen CS, Wang Z, Zhang H, Bu X, Zhang X, An L, Zhang S, Cao Z, Zhan Q, Yang Y, Cao B, Dai H, Liang L, He J; China Pulmonary Health Study Group. Prevalence and risk factors of chronic obstructive pulmonary disease in China (the China Pulmonary Health [CPH] study): a national cross-sectional study. Lancet. 2018 Apr 28;391(10131):1706-1717. doi: 10.1016/S0140-6736(18)30841-9. Epub 2018 Apr 9. PMID 29650248
- [Background] Zhou Y, Zhong NS, Li X, Chen S, Zheng J, Zhao D, Yao W, Zhi R, Wei L, He B, Zhang X, Yang C, Li Y, Li F, Du J, Gui J, Hu B, Bai C, Huang P, Chen G, Xu Y, Wang C, Liang B, Li Y, Hu G, Tan H, Ye X, Ma X, Chen Y, Hu X, Tian J, Zhu X, Shi Z, Du X, Li M, Liu S, Yu R, Zhao J, Ma Q, Xie C, Li X, Chen T, Lin Y, Zeng L, Ye C, Ye W, Luo X, Zeng L, Yu S, Guan WJ, Ran P. Tiotropium in Early-Stage Chronic Obstructive Pulmonary Disease. N Engl J Med. 2017 Sep 7;377(10):923-935. doi: 10.1056/NEJMoa1700228. PMID 28877027
- [Background] Racanelli AC, Kikkers SA, Choi AMK, Cloonan SM. Autophagy and inflammation in chronic respiratory disease. Autophagy. 2018;14(2):221-232. doi: 10.1080/15548627.2017.1389823. Epub 2018 Feb 8. PMID 29130366
- [Background] Zinellu E, Zinellu A, Fois AG, Fois SS, Piras B, Carru C, Pirina P. Reliability and Usefulness of Different Biomarkers of Oxidative Stress in Chronic Obstructive Pulmonary Disease. Oxid Med Cell Longev. 2020 May 14;2020:4982324. doi: 10.1155/2020/4982324. eCollection 2020. PMID 32509143
- [Background] Tang Y, Cai QH, Wang YJ, Fan SH, Zhang ZF, Xiao MQ, Zhu JY, Wu DM, Lu J, Zheng YL. Protective effect of autophagy on endoplasmic reticulum stress induced apoptosis of alveolar epithelial cells in rat models of COPD. Biosci Rep. 2017 Nov 15;37(6):BSR20170803. doi: 10.1042/BSR20170803. Print 2017 Dec 22. PMID 28963374 (Retraction: PMID 34124752 Biosci Rep. 2021 Jun 25;41(6):)
- [Background] Barnes PJ. Inflammatory mechanisms in patients with chronic obstructive pulmonary disease. J Allergy Clin Immunol. 2016 Jul;138(1):16-27. doi: 10.1016/j.jaci.2016.05.011. Epub 2016 May 27. PMID 27373322
- [Background] Balhara J, Gounni AS. The alveolar macrophages in asthma: a double-edged sword. Mucosal Immunol. 2012 Nov;5(6):605-9. doi: 10.1038/mi.2012.74. Epub 2012 Aug 22. PMID 22910216
- [Background] Dewhurst JA, Lea S, Hardaker E, Dungwa JV, Ravi AK, Singh D. Characterisation of lung macrophage subpopulations in COPD patients and controls. Sci Rep. 2017 Aug 2;7(1):7143. doi: 10.1038/s41598-017-07101-2. PMID 28769058
- [Background] Yao Y, Wang Y, Zhang Z, He L, Zhu J, Zhang M, He X, Cheng Z, Ao Q, Cao Y, Yang P, Su Y, Zhao J, Zhang S, Yu Q, Ning Q, Xiang X, Xiong W, Wang CY, Xu Y. Chop Deficiency Protects Mice Against Bleomycin-induced Pulmonary Fibrosis by Attenuating M2 Macrophage Production. Mol Ther. 2016 May;24(5):915-25. doi: 10.1038/mt.2016.36. Epub 2016 Feb 17. PMID 26883801
- [Background] Zhang L, Wang Y, Wu G, Xiong W, Gu W, Wang CY. Macrophages: friend or foe in idiopathic pulmonary fibrosis? Respir Res. 2018 Sep 6;19(1):170. doi: 10.1186/s12931-018-0864-2. PMID 30189872
- [Background] Lea SR, Reynolds SL, Kaur M, Simpson KD, Hall SR, Hessel EM, Singh D. The effects of repeated Toll-like receptors 2 and 4 stimulation in COPD alveolar macrophages. Int J Chron Obstruct Pulmon Dis. 2018 Mar 2;13:771-780. doi: 10.2147/COPD.S97071. eCollection 2018. PMID 29535517
- [Background] Arora S, Dev K, Agarwal B, Das P, Syed MA. Macrophages: Their role, activation and polarization in pulmonary diseases. Immunobiology. 2018 Apr-May;223(4-5):383-396. doi: 10.1016/j.imbio.2017.11.001. Epub 2017 Nov 12. PMID 29146235
- [Background] Zhu YP, Brown JR, Sag D, Zhang L, Suttles J. Adenosine 5'-monophosphate-activated protein kinase regulates IL-10-mediated anti-inflammatory signaling pathways in macrophages. J Immunol. 2015 Jan 15;194(2):584-94. doi: 10.4049/jimmunol.1401024. Epub 2014 Dec 15. PMID 25512602
- [Background] Kunz LI, Lapperre TS, Snoeck-Stroband JB, Budulac SE, Timens W, van Wijngaarden S, Schrumpf JA, Rabe KF, Postma DS, Sterk PJ, Hiemstra PS; Groningen Leiden Universities Corticosteroids in Obstructive Lung Disease Study Group. Smoking status and anti-inflammatory macrophages in bronchoalveolar lavage and induced sputum in COPD. Respir Res. 2011 Mar 22;12(1):34. doi: 10.1186/1465-9921-12-34. PMID 21426578
- [Background] Cornwell WD, Kim V, Fan X, Vega ME, Ramsey FV, Criner GJ, Rogers TJ. Activation and polarization of circulating monocytes in severe chronic obstructive pulmonary disease. BMC Pulm Med. 2018 Jun 15;18(1):101. doi: 10.1186/s12890-018-0664-y. PMID 29907106
- [Background] Kim H, Wang SY, Kwak G, Yang Y, Kwon IC, Kim SH. Exosome-Guided Phenotypic Switch of M1 to M2 Macrophages for Cutaneous Wound Healing. Adv Sci (Weinh). 2019 Aug 27;6(20):1900513. doi: 10.1002/advs.201900513. eCollection 2019 Oct 16. PMID 31637157
- [Background] Fu X, Chen Y, Chen D. The Role of Gut Microbiome in Autoimmune Uveitis. Ophthalmic Res. 2021;64(2):168-177. doi: 10.1159/000510212. Epub 2020 Jul 16. PMID 32674100
- [Background] Martinez FJ, Han MK, Allinson JP, Barr RG, Boucher RC, Calverley PMA, Celli BR, Christenson SA, Crystal RG, Fageras M, Freeman CM, Groenke L, Hoffman EA, Kesimer M, Kostikas K, Paine R 3rd, Rafii S, Rennard SI, Segal LN, Shaykhiev R, Stevenson C, Tal-Singer R, Vestbo J, Woodruff PG, Curtis JL, Wedzicha JA. At the Root: Defining and Halting Progression of Early Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2018 Jun 15;197(12):1540-1551. doi: 10.1164/rccm.201710-2028PP. No abstract available. PMID 29406779
- [Result] Haldar K, George L, Wang Z, Mistry V, Ramsheh MY, Free RC, John C, Reeve NF, Miller BE, Tal-Singer R, Webb AJ, Brookes AJ, Tobin MD, Singh D, Donaldson GC, Wedzicha JA, Brown JR, Barer MR, Brightling CE. The sputum microbiome is distinct between COPD and health, independent of smoking history. Respir Res. 2020 Jul 14;21(1):183. doi: 10.1186/s12931-020-01448-3. PMID 32664956
- [Result] Lopez Caro JC, Santibanez M, Garcia Rivero JL, Villanueva M, Sainz J, Gonzalez Astorqui P, Hierro M, Rodriguez Porres M, Paras Bravo P, Mira A, Rodriguez JC, Galiana A; on behalf of the ACINAR-microbiome study group. Sputum Microbiome Dynamics in Chronic Obstructive Pulmonary Disease Patients during an Exacerbation Event and Post-Stabilization. Respiration. 2019;98(5):447-454. doi: 10.1159/000501988. Epub 2019 Aug 22. PMID 31437842
- [Result] Leitao Filho FS, Alotaibi NM, Ngan D, Tam S, Yang J, Hollander Z, Chen V, FitzGerald JM, Nislow C, Leung JM, Man SFP, Sin DD. Sputum Microbiome Is Associated with 1-Year Mortality after Chronic Obstructive Pulmonary Disease Hospitalizations. Am J Respir Crit Care Med. 2019 May 15;199(10):1205-1213. doi: 10.1164/rccm.201806-1135OC. PMID 30376356